CLINICAL TRIAL: NCT04186910
Title: Increasing Physical Activity in Recovered Persons With Multiple Sclerosis Through Daily Sensor Based Feedback and Weekly Focus Group Meetings: A Feasibility and Pilot II Study
Brief Title: In Clinic Physical Activity in Persons With Multiple Sclerosis
Acronym: PAMS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Physical Activity MS
Record Dates: First submitted 2019-07-04; First posted 2019-12-05 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-07

CONDITIONS: Rehabilitation; Multiple Sclerosis
Keywords: Multiple Sclerosis; Physical activity; Mobility; Self efficacy
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Two arms interventional single blind pilot study
Who Masked: Outcomes Assessor
Masking Description: Assessor will be blind to participants' intervention assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): The control group will not receive any feedback on levels of physical activities but will receive any planned usual care rehabilitation activities
  Interventions: Behavioral: Control group
- Feedback group (Experimental): The feedback group will have an active feedback intervention of physical activities, consisted of daily feedback, received through a Fitbit application, and weekly meeting group focused on enhancing behavioral strategies to increase self-efficacy and motivation. The experimental group will receive any planned usual care rehabilitation activities.
  Interventions: Behavioral: Feedback group

INTERVENTIONS:
Behavioral: Control group — The control group will carry the Fitbit for the entire period of the recovery but will receive no feedback and will not have the app downloaded onto the telephone.
  Arms: Control group
Behavioral: Feedback group — The feedback group will carry the Fitbit for the entire period of the recovery and will receive daily feedback on amount of physical activity carried out and percentage completed of target behavior at the end of the day from an app downloaded on their telephone. The feedback group will also participate in weekly one hour meetings focused on enhancing behavioral strategies to increase self-efficacy and motivation. They will also have their fitbit data analyzed and an agreed upon target of daily activity level increase.
  Arms: Feedback group

SUMMARY:
The aim of htis study is to investigate the post intervention effects of daily feedback on actual physical activity levels derived from a wristworn accelerometer FITBIT combined with self-management training on in-clinic physical activity in persons with moderate to severe disability from MS.

DETAILED DESCRIPTION:
Evidence from various sources indicate that physical activities and mobility practice are beneficial to maintain or increase functional levels in persons with Multiple sclerosis. Even so persons with moderate and severe disability from Multiple sclerosis are less active in daily life than their healthy counterparts. Also during hospital stay persons with MS tend to remain relatively sedentary outside of their rehabilitation sessions. Feedback about physical activity enabled by wearable sensors combined with behavioral strategies to improve self-efficacy and motivation are potential method increase physical activity in hospital inpatients. The primary purpose of this feasibility and interventional study was to determine whether a minimalist physical activity tracker-based feedback and self efficacy training would lead to an increase in physical activity, mobility and quality of life measures during recovery in a group of persons with MS compared to a control group that does not receive feedback. Secondary purpose was to verify if this intervention during recovery would lead to increased perceived physical activity in daily home life after discharge and over longer periods (Follow up at 6 weeks). The study participants will be 60 persons that have moderate to severe disability due to MS, that are admitted to MS Centre of the Santa Maria Nascente Institute, Don Gnocchi Foundation (Milan, Italy). Participants will all receive standard rehabilitation offered in the center. All participants will wear the accelerometer device (FitBit Charge tracker, FitBit Inc, CA, USA) 24 hours per day in order to measure physical activity levels during their hospital stay (3-4 weeks. The participants will be randomized to a group that has no feedback of physical activity level and a group that will have an active feedback intervention (AF). The active feedback intervention will consist of daily feedback, received through a Fitbit application downloaded on their telephones, on whether or not their target activity level was met and how far they were from the target. Additionally, the participants will participate in weekly meeting group focused on enhancing behavioral strategies to increase self-efficacy and motivation. Covariates such as age, sex, stage of change for physical activity behavior, clinical mobility, fatigue, health perception and goal commitment will be measured in all 60 participants both pre and post the intervention/hospital recovery period. The long-term effects on daily perceived functional mobility and self-efficacy will be investigated six weeks after discharge through questionnaires during a telephone call.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MS according to the McDonald's criteria McDonald Criteria 2010
* EDSS score >4.5-7
* Freedom from relapses and steroid treatment for at least 1 month
* Ability to walk at least 10 meters independently with or without support
* MS without relapses in the last 3 months

Exclusion Criteria:

* Mini Mental State Examination (MMSE) score < 20
* The presence of disabling pain or severe deficit of visual acuity
* The presence of severe deficit in communication and severe dysmetry

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Number of passes with Fitbit wristband | Change from number of passes at baseline to number of passes after 4 weeks will be measured.
  A Fitbit wristband consists of an accelerometer and a memory unit and is used to collect mobility data, in the form of number of passes. More passes carried out during the period of wearing the wristband the better.
The 2 minute walking test | Change on the measue will be measured. Will be applied at Day 1 and after 4 weeks
  The 2 minute walking test is used to understand functional mobility. A smaller distance covered (in meters) represents a worse outcome.
The Self-Efficacy in Multiple Sclerosis Scale | Change on the measure will be measured. Will be applied at Day 1, after 4 weeks and after 10 weeks
  The Self-Efficacy in Multiple Sclerosis Scale is a questionnaire of perceived self-efficacy of MS patients

SECONDARY OUTCOMES:
The 10 meters walking scale | Change from Day 1 to day 28 will be measured. Will be applied at the Day 1 and after 4 weeks
  The 10 meters walking test (10MWT) is a test in which the participant is timed while walking 10m at their comfortable speed. A lower gait velocity represents a worse outcome.
The Short Form-12 questionnaire | Change from Day 1 to 4 weeks and until 10 weeks will be measured. Will be applied at baseline Day 1 after 4 weeks and after 10 weeks
  The Short Form-12 questionnaire is comprised of two domains, physical and mental and gives two composite scores that reflect the perceived health of the participant (normative score value= 50).
The EQ-5D visual analogue scale | Change from Day 1 to 4 weeks and until 10 weeks will be measured. Will be applied at the Day 1, after 4 weeks and after 10 weeks
  The EQ-5D visual analogue scale is a measure of health-related quality of life (Minimum score=5, maximum score= 25; higher values represent a worse outcome).
The Twelve Item MS Walking Scale | Change from Day 1 to 4 weeks and until 10 weeks will be measured. Will be applied at the Day 1, after 4 weeks and after 10 weeks
  The Twelve Item MS Walking Scale is a questionnaire about the ability to walk (Minimum score=12, maximum score= 60; higher values represent a worse outcome).
The Fatigue severity Scale | Change from Day 1 to 4 weeks and until 10 weeks will be measured. Will be applied at the Day 1, after 4 weeks and after 10 weeks
  The Fatigue severity Scale is a questionnaire of perception of fatigue (Minimum score=9, maximum score= 63; higher values represent a worse outcome).
The Physical Activity Disability Survey-Revised questionnaire | Change from Day 1 to 4 weeks and until 10 weeks will be measured. Will be applied at the Day 1, after 4 weeks and after 10 weeks
  The Physical Activity Disability Survey-Revised is a questionnaire of physical activity

CONTACTS AND LOCATIONS:
Overall Officials: Johanna Jonsdottir, PhD, Principal Investigator — Senior researcher; Gloria Perini, MSc, Study Director — Researcher
Locations (1):
- Fondazione Don Carlo Gnocchi IRCCS, Milan, Italy

IPD SHARING:
Plan to Share IPD: No
Due to ethical restrictions set by the Ethics Committee of Fondazione Don Carlo Gnocchi and the presence of identifying patient information, researchers wishing to access raw data for use in future research studies should write to the Corresponding Author/Principal investigator that will apply to the Ethics Committee of Fondazione Don Carlo Gnocchi for approval. Additional data can be made available upon request.